CLINICAL TRIAL: NCT06022471
Title: Outcome of Stapes Surgery in Otosclerotic Patients With Tinnitus
Brief Title: Outcome of Stapes Surgery in Otosclerotic Patients With Tinnitus Using Tinnitogram
Acronym: Otosclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Araby Mohamed, Resident doctor at Otolaryngology Departement, Principal Investigator, Assiut University
Other Study IDs: Outcome of ss in ot
Record Dates: First submitted 2023-07-25; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-07

CONDITIONS: Otosclerosis
MeSH Terms: conditions — Otosclerosis | interventions — Stapes Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stapes surgery
  Interventions: Procedure: Stapes surgery

INTERVENTIONS:
Procedure: Stapes surgery — Stapedectomy operation

SUMMARY:
This study will be conducted on patients with otosclerosis attending Assiut University Hospital and undergo stapedectomy operation Evaluation of each patient will conducted preoperatively and 3 month postoperatively Patient will undergo tinnitogram and tinnitus handicap questionnaire before and after the operation to measure improvement in hearing and tinnitus

DETAILED DESCRIPTION:
Otosclerosis is an abnormal bone remodeling in the middle ear The normal dense endochondral layer of the bony otic capsule in the labyrinth is replaced by irregularly laid spongy bone leading to the fixation of the stapes.

* Clinical otosclerosis is more prevalent in females than in males, giving rise to the hypothesis that sex hormones may contribute to the development of disease
* The age of onset is variable, although hearing loss typically begins in the third decade, with a range from first decade to the sixth decade.

In most cases, hearing loss is bilateral (70-85%) and is usually asymmetrical, developing initially in one ear before progressing to the other.

Positive family history of otosclerosis has been previously reported in between 30-70% of cases.

The diagnosis is usually made clinically by

* History
* Physical examination,
* Audiogram results(tinnitus handicap questionnaire arabic version, tinnnitogram ) most frequent presentation of patients with clinical otosclerosis is bilateral hearing loss and tinnitus Between 65 and 87% of patient with otosclerosis experience tinnitus. most of them has unilateral tinnitus 83.3% , while only 16.7% reported bilateral tinnitus.

patients with tinnitus often report that their tinnitus is associated with feelings of sadness, worry, frustration, and anger.

These feelings can lead to difficulties sleeping, relaxing, and concentrating and may negatively impact relationships at work and impair participation in social settings .

Stapedotomy through sufficient air-bone gap closure Data collection

1. full history taking
2. tinnitus handicap questionnaire arabic version
3. Vital signs and general examination
4. Full ENT examination including ear canal and tympanic membrane examination
5. Routine audiologic testing which provide an assessment of patient hearing
6. Investigation
7. Preoperative fitness
8. Tinnitogra

Tinnitogram :

Tinnitus pitch match : we will start at 1000 Hz and move up and down in frequency.

Tinnitus loudness match : patient threshold was determined at frequency of pitch matching, sound level will increase in small steps(1or 2 dB ) until patient repoted that specific tone will just equal in loudeness to his tinnitus Tinnitus handicap questionnaire arabic version

ELIGIBILITY:
Inclusion Criteria:

* patient with otosclerosis undergo stapes surgery in otorhinology department in Assiut university hospital
* All patient have tinnitus and conductive hearing loss or mixed hearing loss.

Exclusion Criteria:

* patient with otosclerosis who don't undergo stapes surgery patient have tinnitus due to causes other than otosclerosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patient with conductive hearing loss associated with tinnitus
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
decrease tinnitus | 3 month
  Measuring tinnitus by tinnitogram By pure tone averages untile patients report that specific tone resemble their tinnitus The unit of measure for sound intensity is the decibel (dB)

SECONDARY OUTCOMES:
Changes in pure tone averages | 3 month
  Pure tone averages calculated from pure tone audiometry will be summarized using the mean

IPD SHARING:
Plan to Share IPD: No